CLINICAL TRIAL: NCT00914290
Title: A Study With IPX056 in Subjects With Spasticity Associated With Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Impax Laboratories, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IPX056-B09-01
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2017-05

CONDITIONS: Spasticity; Multiple Sclerosis
MeSH Terms: conditions — Muscle Spasticity; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IPX056-Baclofen IR-IPX056 (Other): Following 2 weeks of run-in period, subjects were randomized to IPX056 and Placebo IR for 2 weeks and then to Baclofen IR and Placebo IPX056 for 2 weeks.
  Interventions: Drug: IPX056; Drug: Baclofen IR; Drug: Placebo IPX056; Drug: Placebo IR
- IPX056-IPX056-Baclofen IR (Active Comparator): Following 2 weeks of run-in period, subjects were randomized to Baclofen IR and Placebo IPX056 for 2 weeks and then to IPX056 and Placebo IR for 2 weeks.
  Interventions: Drug: IPX056; Drug: Baclofen IR; Drug: Placebo IPX056; Drug: Placebo IR

INTERVENTIONS:
Drug: IPX056 — IPX056 ER capsule containing 10 mg baclofen
  Other Names: IPX056 ER Capsule; IPX056 ER
Drug: Baclofen IR — Encapsulated baclofen tablet 5 mg per capsule
  Other Names: CAS Registry Number [11134-47-0]
Drug: Placebo IPX056 — Placebo capsule for IPX056
Drug: Placebo IR — Placebo encapsulated baclofen placebo tablet

SUMMARY:
To explore the safety and efficacy of IPX056 compared with baclofen tablets for alleviation of symptoms of spasticity associated with multiple sclerosis (MS).

DETAILED DESCRIPTION:
IPX056 was compared with commercially available tablets as it was designed to provide a prolonged duration of absorption to reduce dose frequency and/or to provide prolonged duration of antispasticity effect.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years old.
* Agrees to use a medically acceptable method of contraception throughout the study
* Diagnosed with MS as defined by Poser or McDonald Criteria.
* Receiving commercial baclofen tablets at a stable total daily dose ranging from 15 mg to 80 mg in a TID dosing regimen for at least 4 weeks prior to the Screening Visit that has resulted in improved spasticity.
* Willing to wash out and remain off other antispasticity medications during the study.

Exclusion Criteria:

* If female, the subject is pregnant, planning to become pregnant, or breastfeeding.
* History of allergy or severe intolerance to baclofen.
* Did not respond to previous baclofen treatment in any formulation.
* Has experienced an exacerbation of MS within 1 month.
* Urinary tract infection (UTI) within 2 weeks or two symptomatic UTIs within 6 months prior to the study.
* Subjects with clinically significant impairment of renal function
* History of active seizure disorder or epilepsy, or currently taking an anticonvulsant for treatment or control of seizure.
* Other conditions causing spasticity (e.g., stroke, cerebral palsy, traumatic brain injury) or rigidity (e.g. Parkinson's Disease).
* Treated with Botulinum Toxin Type A or B within the previous 4 months, or with phenol or therapeutic alcohol nerve block within 12 months or planned use of these drugs during this study.
* Has clinically significant limitation of passive range of motion of lower extremities.
* Has had major surgery within 6 months prior to Screening Visit that may affect spasticity assessments such as abdominal surgery, back surgery, lower leg and knee surgeries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-04; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Morning Stiffness Score | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Impax Study Director, Study Director — Impax Laboratories, LLC
Locations (11):
- United States (11):
  - Northwest NeuroSpecialists, PLLC, Tucson, Arizona
  - University of Colorado, Aurora, Colorado
  - Meridien Research, Tampa, Florida
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - MidAmerica Neuroscience Institute, Lenexa, Kansas
  - QUEST Research Institute, Bingham Farms, Michigan
  - Great Falls Cllinic, Great Falls, Montana
  - Empire Neurology, PC, Latham, New York
  - Winthrop University Hospital, Mineola, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Central Texas Neurology Consultants, Round Rock, Texas

IPD SHARING:
Plan to Share IPD: No